CLINICAL TRIAL: NCT02982005
Title: A Phase 3 Multicenter, Randomized, Double-blind, Placebo-controlled Study With an Open Label Extension to Evaluate the Efficacy and Safety of KHK4827 in Subjects With Moderate to Severe Plaque Psoriasis
Brief Title: A Study of KHK4827 (Brodalumab) in Subjects With Moderate to Severe Psoriasis in Korea
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Kyowa Kirin Korea Co., Ltd. (Industry)
Responsible Party: Sponsor
Organization: Kyowa Kirin Co., Ltd. (Industry)
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 4827-KR001
Record Dates: First submitted 2016-12-01; First posted 2016-12-05 (Estimated); Last update posted 2024-04-29 (Actual); Status verified 2024-04

CONDITIONS: Moderate to Severe Plaque Psoriasis
Keywords: KHK4827 (brodalumab)
MeSH Terms: interventions — brodalumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- KHK4827 (Experimental): KHK4827 administered SC
  Interventions: Drug: KHK4827
- Placebo (Placebo Comparator): Placebo administered SC
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: KHK4827 — Administered KHK4827 by subcutaneous (SC) injection until week 62.
  Other Names: Brodalumab
  Arms: KHK4827
Drug: Placebo — Administered placebo by subcutaneous (SC) injection until week 12. Administered KHK4827 by SC injection from week 13 until week 62.
  Arms: Placebo

SUMMARY:
The primary objective of this study is to evaluate the efficacy and safety of KHK4827 in subjects with moderate to severe plaque psoriasis randomized in a double-blind manner to receive KHK4827 or placebo for 12 weeks

ELIGIBILITY:
Inclusion Criteria:

* Subject has had stable moderate to severe plaque psoriasis for at least 6 months
* Subject has involved BSA ≧ 10%, PASI ≧ 12, and sPGA ≧ 3 at screening and at baseline

Exclusion Criteria:

* Subject diagnosed with erythrodermic psoriasis, pustular psoriasis, guttate psoriasis, or a medication-induced psoriasis, or other skin conditions (e.g., eczema) at screening that would interfere with study evaluations
* Subject scheduled to undergo a surgical intervention during the study period
* Subject has any active infection or history of infections as defined in the study protocol
* Subject has known history of Crohn's disease
* Subject has any other significant concurrent medical condition or laboratory abnormalities, as defined in the study protocol
* Subject has not stopped using certain psoriasis therapies as defined in the study protocol
* Subject has previously used any anti-IL-17 biologic therapy
* Subject is pregnant or breast feeding, or planning to become pregnant while enrolled in the study
* Women of child-bearing potential or fertile men who do not agree to use effective contraception from the day of providing consent through 12 weeks after the last dose of investigational product.
* Subject has known history or evidence of suicidal ideation (severity of 4 or 5) or any suicidal behavior based on an assessment with the Columbia-Suicide Severity Rating Scale (C-SSRS) at screening or at baseline
* Subject has severe depression based on a total score of ≥ 15 on the Patient Health Questionnaire-8 (PHQ-8) at screening or at baseline
* Subject has known history or evidence of a psychiatric disorder that, in the opinion of the investigator, would pose a risk to subject safety or interfere with the study evaluation, procedures or completion
* Subject has known history of alcohol and/or substance abuse within the last 12 months"

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Actual)
Dates: Start 2017-01; Primary Completion 2018-08-14 (Actual); Study Completion 2018-08-14 (Actual)

PRIMARY OUTCOMES:
Psoriasis area and severity index (PASI) 75 response | at week 12
Static physician's global assessment (sPGA) of "0 (clear)" or "1 (almost clear)" | at week 12

SECONDARY OUTCOMES:
PASI 50/75/90/100 response by visit | Baseline to week 64
sPGA of "0 (clear) or 1 (almost clear)" by visit | Baseline to week 64
Body surface area (BSA) involvement of lesion | Baseline to week 64
Nail psoriasis severity index (NAPSI) score (applicable only to subjects who had nail symptoms at baseline) | Baseline to week 64
Psoriasis scalp severity index (PSSI) score (applicable only to subjects who had scalp symptoms at baseline) | Baseline to week 64
Dermatology life quality index (DLQI) | Baseline to week 64
Treatment-emergent adverse events (TEAEs) or drug-related TEAEs | Baseline to week 64
Laboratory values | Baseline to week 64
Vital signs | Baseline to week 64
Anti-KHK4827 antibodies | Baseline, Week 12, Week 24, Week 48, Week 64
Serum KHK4827 concentration | Baseline, Week 8, Week 10, Week 12, Week 24

CONTACTS AND LOCATIONS:
Locations (1):
- Korea, Republic of, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No